CLINICAL TRIAL: NCT04998383
Title: HVNI vs Noninvasive Ventilation for Acute Hypercapnic Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nagah Gaber, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HVNI
Record Dates: First submitted 2021-08-02; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Comparison Between HVNI vs Noninvasive Ventilation for Acute Hypercapnic Respiratory Failure

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either high-velocity nasal insufflation or noninvasive positive-pressure ventilation therapy and they will be enrolled if they met the inclusion criteria.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HVNI (Experimental): High velocity nasal insufflation (Fisher &Paykel, Auckland, New Zealan High-velocity nasal insufflation (Precision Flow;Vapotherm, Inc, Exeter, NH) (Figure 2) using a smallborenasal cannula was initiated with a flow rate set to 35 L/min, with a starting temperature between 35C and 37C and FiO2 at 1.0. Adjustments in flow (up to 40 L/min) and temperature (typically between 35C and 37C) were made to alleviate respiratory distress and optimize comfort
  Interventions: Device: HVNI
- Noninvasive ventilation (Experimental): Respiratory assistance is provided by a NIV either Puritan Bennet 840 (Covidien, U.S.A.), EngströmCarestation (GE Healthcare, Finland) or Hamilton-G5 (Hamilton Medical, Germany), will be used for conventional non-invasive ventilation via an oronasal mask that helps patients to cope with their Breathlessness. Settings will be adjusted based on the clinical assessment of the respiratory therapist as per standard practice.
  Interventions: Device: HVNI

INTERVENTIONS:
Device: HVNI — High velocity nasal insufflation (Fisher &Paykel, Auckland, New Zealan High-velocity nasal insufflation (Precision Flow;Vapotherm, Inc, Exeter, NH) (Figure 2) using a smallborenasal cannula was initiated with a flow rate set to 35 L/min, with a starting temperature between 35C and 37C and FiO2 at 1.0. Adjustments in flow (up to 40 L/min) and temperature (typically between 35C and 37C) were made to alleviate respiratory distress and optimize comfort.

SUMMARY:
1. To study the efficacy and safety of high flow nasal oxygenation using high velocity nasal insfflation technique(HiVNI) in comarison with non invasive positive pressure ventilation in COPD patients with acute hyercapnic respiratory failure
2. To do selection criteria for the indication of this new physiological technique in critically ill COPD patients

DETAILED DESCRIPTION:
Dyspnea and acute respiratory failure are among the top 5 reasons for patients to present to the emergency department (ED)(1).Supplemental oxygen therapy forms the cornerstone of resuscitation of the acutely unwell patient.Under normal circumstances, tissue hypoxia occurs within 4 min of inadequate tissue oxygenation (2). Oxygen delivery to the peripheral tissues depends upon the product of cardiac output and the arterial oxygen content (3), which is partly dependent on FIO2. In intensive care unit (ICU) patients with acute respiratory failure, non-invasive strategies of oxygenation are mainly used to avoid invasive mechanical ventilation (4). In such situations, the goal of treatment should not only be survival, but also improved respiratory condition and avoidance of inappropriate discomforts. Since the 90's, noninvasive ventilation (NIV) has been largely used with strong level of evidence in cardiogenic pulmonary edema and chronic obstructive pulmonary disease (COPD) exacerbation. NIV improves gas exchange and reduces inspiratory effort through positive pressure. However, good tolerance to NIV is sometimes difficult to achieve due to frequent leaks around the mask, possibly leading to patientventilator asynchrony and even to intubation. It may have other deleterious effects such as delayed intubation by masking signs of respiratory distress, or barotrauma by the high tidal volume potentially generated under positive pressure (5). High-velocity nasal insufflation (Hi-VNI), a viable alternative to NiPPV in treating adults in undifferentiated respiratory distress. It provides both oxygenation and ventilatory support to reduce hypercapnia(6).It focuses on optimum efficiency of the deadspace purge to augment ventilation (7,8), in addition to delivering up to 100% oxygen by nasal cannula(9,10) This is accomplished by use of small-bore nasal cannulae (typically 2.7-mm internal diameter for adult patients) to produce high velocity flow that is approximately 360% greater than that of the larger bore cannulae. It requires a flow of 25 to 35 L/min in adults to accomplish a complete purge of the extrathoracic anatomic reservoir between breaths (8,11).

ELIGIBILITY:
Inclusion Criteria:Participants admitted to the RICU with acute hypercapnic respiratory failure requiring NIV support with the following criteria:

1. RR> 25 breath/minute.
2. Use of accessory muscles of respiration, paradoxical breathing, thoracoabdominal asynchrony.
3. Hypoxemia evidenced by the following items:

   * In patient with hypercapnic ARF:

I.Need for oxygen therapy at FIO2> 40% to maintain PaO2 > 60 mmHg or SaO2> 90% II.Blood gas analysis shows pH <7.35 and paCO2> 45 mmHg

-

Exclusion Criteria:Patients with ARF who have any of the following:

I.Indication for emergency endotracheal intubation. II.HR < 50 beat\minute with decreased level of consciousness III.Persistent hemodynamic instability with

* Systolic blood pressure <90 mmHg after infusing a bolus of crystalloid solution at a dose of 30 ml / kg.
* life-threatening arrhythmia. IV.Undrained pneumothorax or Pneumothorax with persistent air leak. V.Extensive facial trauma or burnVI.Refusal to participate. VII.Usual long-term treatment with NIV for chronic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Endotracheal intubation rate | after 2 Hours
  Endotracheal intubation rate

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed hamed, prof.dr, Study Director — Assiut University; Khalid Hussein, prof.dr, Study Director — Assiut University; Samiaa Hamdy, assistant professor, Study Director — Assiut University

REFERENCES:
- [Result] Weiss AJ, Wier LM, Stocks C, Blanchard J. Overview of Emergency Department Visits in the United States, 2011. 2014 Jun. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #174. Available from http://www.ncbi.nlm.nih.gov/books/NBK235856/ PMID 25144109
- [Result] Bateman NT, Leach RM. ABC of oxygen. Acute oxygen therapy. BMJ. 1998 Sep 19;317(7161):798-801. doi: 10.1136/bmj.317.7161.798. No abstract available. PMID 9740573
- [Result] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265
- [Result] Frat JP, Coudroy R, Marjanovic N, Thille AW. High-flow nasal oxygen therapy and noninvasive ventilation in the management of acute hypoxemic respiratory failure. Ann Transl Med. 2017 Jul;5(14):297. doi: 10.21037/atm.2017.06.52. PMID 28828372
- [Result] Doshi P, Whittle JS, Bublewicz M, Kearney J, Ashe T, Graham R, Salazar S, Ellis TW Jr, Maynard D, Dennis R, Tillotson A, Hill M, Granado M, Gordon N, Dunlap C, Spivey S, Miller TL. High-Velocity Nasal Insufflation in the Treatment of Respiratory Failure: A Randomized Clinical Trial. Ann Emerg Med. 2018 Jul;72(1):73-83.e5. doi: 10.1016/j.annemergmed.2017.12.006. Epub 2018 Jan 6. PMID 29310868
- [Result] Frizzola M, Miller TL, Rodriguez ME, Zhu Y, Rojas J, Hesek A, Stump A, Shaffer TH, Dysart K. High-flow nasal cannula: impact on oxygenation and ventilation in an acute lung injury model. Pediatr Pulmonol. 2011 Jan;46(1):67-74. doi: 10.1002/ppul.21326. Epub 2010 Nov 23. PMID 21171186
- [Result] Dysart K, Miller TL, Wolfson MR, Shaffer TH. Research in high flow therapy: mechanisms of action. Respir Med. 2009 Oct;103(10):1400-5. doi: 10.1016/j.rmed.2009.04.007. Epub 2009 May 21. PMID 19467849
- [Result] Spoletini G, Alotaibi M, Blasi F, Hill NS. Heated Humidified High-Flow Nasal Oxygen in Adults: Mechanisms of Action and Clinical Implications. Chest. 2015 Jul;148(1):253-261. doi: 10.1378/chest.14-2871. PMID 25742321
- [Result] Mehta S, Jay GD, Woolard RH, Hipona RA, Connolly EM, Cimini DM, Drinkwine JH, Hill NS. Randomized, prospective trial of bilevel versus continuous positive airway pressure in acute pulmonary edema. Crit Care Med. 1997 Apr;25(4):620-8. doi: 10.1097/00003246-199704000-00011. PMID 9142026
- [Result] Tan D, Walline JH, Ling B, Xu Y, Sun J, Wang B, Shan X, Wang Y, Cao P, Zhu Q, Geng P, Xu J. High-flow nasal cannula oxygen therapy versus non-invasive ventilation for chronic obstructive pulmonary disease patients after extubation: a multicenter, randomized controlled trial. Crit Care. 2020 Aug 6;24(1):489. doi: 10.1186/s13054-020-03214-9. PMID 32762701
- [Result] Patrick W, Webster K, Ludwig L, Roberts D, Wiebe P, Younes M. Noninvasive positive-pressure ventilation in acute respiratory distress without prior chronic respiratory failure. Am J Respir Crit Care Med. 1996 Mar;153(3):1005-11. doi: 10.1164/ajrccm.153.3.8630538.